CLINICAL TRIAL: NCT01091987
Title: Pilot Study on the Feasibility of Non-pharmacological Treatment of Insomnia in Nursing Homes.
Brief Title: Non-pharmacological Treatment of Insomnia in Nursing Homes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Flemish Minister for Welfare, Public Health and Family, Belgium (Unknown); Farmaka vzw, Belgium (Unknown); Domus Medica vzw, Belgium (Unknown)
Responsible Party: Thierry Christiaens, MD, PhD, University Ghent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010/031
Record Dates: First submitted 2010-03-19; First posted 2010-03-24 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Insomnia
Keywords: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Non-pharmacological approach of insomnia (Experimental): Non-pharmacological approach of insomnia based on cognitive-behavioural techniques (education on sleep, sleep hygiene, stimulus control, cognitive techniques)
  Interventions: Behavioral: Non-pharmacological approach of insomnia

INTERVENTIONS:
Behavioral: Non-pharmacological approach of insomnia — education on sleep, sleep hygiene, stimulus control, cognitive techniques

SUMMARY:
The study wants to examine the feasibility of a non-pharmacological approach for insomnia in nursing homes provided by trained nurses/paramedics and physicians.

ELIGIBILITY:
Inclusion Criteria:

* Male and female nursing home residents of age 55+ with insomnia, defined as difficulty in getting to sleep, difficulty in staying asleep, early wakening, or non-restorative sleep

Exclusion Criteria:

* insufficient cognitive ability for self-reflection
* dementia
* insomnia caused by a medical disorder (hyperthyroidism, congestive heart failure, peripheral arterial disease, GORD, COPD/asthma, angina pectoris, benign prostatic hyperplasia, arthritis, other
* insomnia caused by medication
* substance misuse
* other sleep disorder: restless legs syndrome, periodic limb movement disorder, sleep apnoea, narcolepsy
* psychiatric disorder: psychotic or bipolar disorder in anamnesis, major depression present or more than 2 episodes in anamnesis
* short stay

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The proportion of eligible residents who accepted to participate in the non-pharmacological program and the proportion of eligible residents who completed the non-pharmacological program. | after 3 months
  Evaluation takes place at the moment the program is ended according to the trained caregiver or maximally 3 months after the start of the program.

SECONDARY OUTCOMES:
Insomnia, as measured by the Groningen Sleep Quality Questionnaire | at baseline and after 3 months
quality of life | at baseline and after 3 months
  measured by the Geriatric Behaviour Observation Scale
Use of sleep medication | at baseline and after 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Christiaens, MD, PhD, Principal Investigator — University Ghent
Locations (1):
- University Ghent, Ghent, Belgium